CLINICAL TRIAL: NCT05787054
Title: Single Scan Screening of Fetal Growth Restriction Versus Longitudinal Scan Screening in the Third Trimester: a Multicenter Randomized Protocol
Brief Title: Third Trimester Screening of Fetal Growth Restriction
Acronym: RELAIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 1909
Record Dates: First submitted 2023-02-21; First posted 2023-03-28 (Actual); Results first posted 2025-04-30 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2023-05

CONDITIONS: Fetal Growth Retardation; Fetal; Slow Growth
MeSH Terms: conditions — Fetal Growth Retardation

STUDY DESIGN:
Intervention Model Description: 1:1
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single scan (Active Comparator): Single scan at 28-32 weeks
  Interventions: Other: Third trimester ultrasound
- Longitudinal scan (Experimental): Longitudinal scan at 28-32 AND 35-37 weeks
  Interventions: Other: Third trimester ultrasound

INTERVENTIONS:
Other: Third trimester ultrasound — Single scan versus Longitudinal scan

SUMMARY:
The aim of this trial is to assess the efficacy of two screening protocols for the detection of fetal growth disorders.

In Italy at the moment the screening protocol should not be universal but only on clinical indications. In some Regions the screening is offered to every pregnant women with an early third trimester scan at 28-32 weeks'gestation or, in other Regions, according to the new national recommandations, a growth scan during the third trimester is provided only if there is a clinical indication.

DETAILED DESCRIPTION:
The Aim of this trial is to assess the efficacy and efficiency of two screening protocols for fetal growth disorders: one providing an early fetal growth assessment at 28-32 weeks' (single scan) and the second one with the addition of a late third trimester screening at 35-37 weeks (longitudinal scan).

This study is designed to generate level 1 evidence of diagnostic efficacy.

MAIN OUTCOME: The main outcome of the two protocols in screening true late SGA fetuses is measured based on the antenatal detection of small for gestational age newborn basing on the IG21th newborn weight charts centiles <the 10th according to gestational age and gender at delivery.

SECONDARY OUTCOME

* Antenatal detection of severe SGA <3rd centile
* Mode of delivery
* Caesarean section rate according to Robson classes for singleton
* Composite mild adverse neonatal outcome (Apgar score at 5 minutes <7, pH < 7.10, or BD >8mmol/L, admission at NICU)
* Composite severe adverse perinatal (stillbirth or term live birth associated with neonatal death, hypoxic ischaemic encephalopathy, use of inotropes, need for mechanical ventilation, or severe metabolic acidosis (defined as a cord blood pH <7•0 and base deficit >12 mmol/L)

TERTIARY OUTCOME

* Number of ultrasound scans performed in outpatient clinics by medical indication (SSR-prescription) beyond Early-TT and late-TT scheduled exams, and number of ultrasound scans performed on indication in outpatient clinics minus the first one indicated.
* Number of ultrasound scans by patient choice
* Econometrics of the two protocols, and of the estimated sanitary costs of outcomes

4.2 EXPERIMENTAL PLAN

Women who agree to participate are randomized to a single scan Protocol vs longitudinal Scan protocol.

5. STUDY POPULATION

Sample size is based on sensitivity in detecting SGA below 10th centile weight at birth. For the 28-32 group, sensitivity is based on results by Roma et al. (22.5%). The results published by Sovio et al. are instead taken for the "longitudinal" group (57% sensitivity). The sample size calculation was carried out for the comparison between the 28-32 only group vs. the "longitudinal". The calculation considered a confidence level of 95% (1-alpha) and an 80% power (1-beta), and a one to one ratio between the 28-32 only groups and the "longitudinal". According to Fleiss (Fleiss JL. Statistical methodsf or rates and proportions, II Ed. John Wiley & Sons, New York, 1981. page45, formulas 3.18 & 3.19), for the 28-32 only group vs. the "longitudinal",each arm should be 32 women, which implies 64 for two arms. SGA represent, as by definition, 10% of the total population: the sample size needed considering both AGA and SGA, is then 64x10=640. Considering 10% of drop-out and incomplete data the final sample size should be increased of such percentage, reaching 704 subjects. The sample should be recruited according to the number of deliveries per year of each institute involved in the multicenter study.

5.2 PATIENT SELECTION 5.2.1 INCLUSION CRITERIA Eligible cases are nulliparous pregnant women, with first trimester ultrasound assessment of gestational age, who conceived singleton fetuses. If the crown-rump-length (CRL) differs of more than ± 3-5 days from the last menstrual period, gestational age is calculated on the CRL.

5.2.2 EXCLUSION CRITERIA

* major medical disease
* high risk for preeclampsia on history or detected in those centres that perform pre-eclampsia screening at first trimester
* women older than 40 years on ASA low dose prophylaxis
* known immune disorders or clinical thrombophilic conditions;
* twin pregnancies;
* IVF
* suspected fetal anomalies
* Papp-A at Combined-Test<0.2

5.3 WITHDRAWAL PROCEDURES If a patient, during the study protocol, wanted to withdrawal, this will not modify the subsequent monitoring of her pregnancy following local protocols.

6. SUBJECT TREATMENT

• RANDOMIZATION : Patients who agree to participate and sign an informed consent, Women who agree to participate are randomized to the single scan Protocol vs Longitudinal-TT protocols.

ELIGIBILITY:
Inclusion Criteria:

* Eligible cases are nulliparous pregnant women, with first trimester ultrasound assessment of gestational age, who conceived singleton fetuses. If the crown-rump-length (CRL) differs of more than ± 3-5 days from the last menstrual period, gestational age is calculated on the CRL.

Exclusion Criteria:

* major medical disease
* high risk for preeclampsia on history or detected in those centres that perform pre-eclampsia screening at first trimester
* women older than 40 years on ASA low dose prophylaxis
* known immune disorders or clinical thrombophilic conditions;
* twin pregnancies;
* IVF
* suspected fetal anomalies at any gestational age
* Papp-A at Combined-Test<0.2

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — pregnant women
Enrollment: 813 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-05-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alessandra Familiari, MD, Principal Investigator — Catholic University of the Sacred Heart, Rome
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli IRCCS, UOC Ostetricia e Patologia ostetrica, Rome, RM, Italy

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD
Supporting Information: CSR
Time Frame: When the first publication is ready for submission for one year
Access Criteria: Only for principal investigators of the recruiting centres

REFERENCES:
- [Derived] Familiari A, Stampalija T, Prefumo F, di Marco G, Ferrante MG, Bevilacqua E, Zamagni G, Monasta L, Tiralongo G, Valensise H, Morlando M, Sarno L, Di Mascio D, Mappa I, Rizzo G, Visentin S, Fichera A, Radaelli T, Thilaganathan B, Scambia G, Ghi T, Ferrazzi E. Single versus longitudinal scans in the third trimester: a multicenter randomized clinical trial on screening for late-onset intrauterine fetal growth restriction (The RCT on Evaluation of LAte Iugr Screening study). Am J Obstet Gynecol. 2025 Nov 21:S0002-9378(25)00858-0. doi: 10.1016/j.ajog.2025.11.027. Online ahead of print. PMID 41276199

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Single Scan | Longitudinal Scan
Started | 407 | 406
Completed | 396 | 394
Not Completed | 11 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Single Scan | Longitudinal Scan | Total
Number analyzed (Participants) | 396 | 394 | 790
Age, Continuous [Mean (Full Range); unit: years] | 30.7 [18 to 40] | 30.7 [18 to 40] | 30.7 [18 to 40]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 396 | 394 | 790
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 5 | 9
  Not Hispanic or Latino | 390 | 389 | 779
  Unknown or Not Reported | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  Italy | 396 | 394 | 790

OUTCOME MEASURES:

1. Primary Outcome: Rate of Small for Gestational Age at Birth Identified Antenatally
Description: Rate of newborns with a Birth Weight <10 th centile according to International Prescriptive Charts who were prenatally identified
Time Frame: at birth
Population: sensibility of two screening protocols
Measure: Count of Participants; unit: Participants
Arm/Group | Single Scan | Longitudinal Scan
Number analyzed (Participants) | 396 | 394
Participants | 28 | 46

2. Secondary Outcome: Rate of Cesarean Section in the Two Groups
Description: Rate of patients undergoing C section rather than spontaneous vaginal birth
Time Frame: at birth
Population: Odds Ratio for Cesarean section
Measure: Count of Participants; unit: Participants
Arm/Group | Single Scan | Longitudinal Scan
Number analyzed (Participants) | 396 | 394
Participants | 84 | 76

3. Secondary Outcome: Rate of Adverse Outcomes
Description: rate of admission into neonatal intensive care unit
Time Frame: up to 40 days after birth
Population: rate of neonatal admission into intensive care unit
Measure: Count of Participants; unit: Participants
Arm/Group | Single Scan | Longitudinal Scan
Number analyzed (Participants) | 396 | 394
Participants | 15 | 4

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Single Scan | Longitudinal Scan
All-Cause Mortality (participants affected / at risk) | 1/396 | 0/394
Serious Adverse Events (participants affected / at risk) | 0/396 | 0/394
Other Adverse Events (participants affected / at risk) | 0/396 | 0/394

LIMITATIONS AND CAVEATS:
Limitations of our study include that the sample size has been calculated to determine the diagnostic effectiveness of the two screening protocols and not on perinatal outcomes - that represent a secondary outcome - thus meaning that possible additional differences in neonatal outcomes could be shown in a larger population, and we did not explore whether the intervention had any effect on long term consequences

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-19): https://cdn.clinicaltrials.gov/large-docs/54/NCT05787054/Prot_SAP_001.pdf